CLINICAL TRIAL: NCT06309927
Title: Operative Hysteroscopy Versus Suction Curettage for Surgical Termination of Early Pregnancy Loss (Miscarriage)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Noam Smorgick, Director of Minimally Invasive Gynecologic Surgery, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0025-24-ASF
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Early Pregnancy Loss; Intrauterine Adhesion
Keywords: hysteroscopy; curettage; early pregnancy loss; tissue removal device
MeSH Terms: conditions — Abortion, Spontaneous; Gynatresia | interventions — Vacuum Curettage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Operative hysteroscopy (Experimental): Surgical evacuation of the uterine cavity by operative hysteroscopy (tissue removal device, Truclear Mini-Elite)
  Interventions: Procedure: Operative hysteroscopy (by tissue removal device)
- Suction curettage (Active Comparator): Surgical evacuation of the uterine cavity by ultrasound guided suction curettage
  Interventions: Procedure: Suction curettage

INTERVENTIONS:
Procedure: Operative hysteroscopy (by tissue removal device) — Surgical evacuation of the uterine cavity using the Truclear Mini-Elite hysteroscopic tissue removal device
  Arms: Operative hysteroscopy
Procedure: Suction curettage — Surgical evacuation of the uterine cavity with electrical vacuum suction curette
  Arms: Suction curettage

SUMMARY:
Non-blinded prospective randomized study. 100 women diagnosed with early pregnancy loss up to 10 gestational weeks who opted for surgical management (after being offered the options of conservative management and medical treatment) will be recruited.

Qualifying patients will sign an informed consent form and will be randomly assigned to the two arms of the study:

1. Surgical uterine evacuation by the traditional ultrasound-guided suction curettage (control group)
2. Surgical uterine evacuation by operative hysteroscopy using a tissue removal device (study group).

The surgical procedure will be determined randomly by computer generated allocation.

All surgical procedures will be performed under general anesthesia in an outpatient surgical suite. The operative time, operative blood loss and intraoperative complications will be recorded by the research team.

Following the surgical procedure, the patients will be monitored and discharged home as per our department's day-surgery protocol. Immediate post-operative complications will be recorded until discharge.

One week after the procedure, a telephone interview will be conducted to assess any procedure-related complications.

A diagnostic hysteroscopy without anesthesia will be scheduled 6 weeks postoperatively to assess for retained products of conception and for intrauterine adhesions. The diagnostic hysteroscopy will be performed by a practitioner who will be blinded to the type of surgery performed.

6 months after the procedure, a telephone questionnaire will be conducted to assess for subsequent pregnancies.

DETAILED DESCRIPTION:
Early pregnancy loss occurs in ~ 15% of all pregnancies, while 10% of women have experienced at least one pregnancy loss. The therapeutic options that are available in these cases include surgical termination of pregnancy by suction curettage, medical treatment with Misoprostol, and conservative management. The surgical termination of pregnancy allows for relatively quick termination of the pregnancy, and prevention of heavy vaginal bleeding requiring urgent curettage. However, although this is a common and relatively safe procedure, it is associated with risks such as infection, residual trophoblastic tissue or retained products of conception (RPOC), bleeding and uterine perforation. In the long term, there is a risk of intrauterine adhesions formation, which may cause infertility and in severe cases, Asherman's syndrome. It has been hypothesized that RPOC following suction curettage occur because it is a "blind" operation. Therefore, it is now common practice to use ultrasound imaging during and/or immediately after the procedure in order to verify that all the pregnancy contents have been removed. However, despite the use of ultrasound, RPOCs are diagnosed in 1% to 10% of these procedures. Intrauterine adhesions following suction curettage are another significant risk of these procedures. In a study by Hooker et al., intrauterine adhesions were found in approximately 20% of suction curettage cases, while in women with repeated miscarriages the risk of intrauterine adhesions was even higher. Intrauterine adhesions are of critical importance in women of childbearing age, as they may cause infertility, menstrual disorders, and recurrent miscarriages. Therefore, preventing adhesions or reducing the rate of adhesions after surgical emptying of the uterine cavity is an issue of utmost importance in women of childbearing age. Thus, in recent years, several studies have investigated the use of operative hysteroscopy for surgical evacuation of early pregnancy loss. Hysteroscopy allows a visual assessment of the uterine cavity (as opposed to a "blind" suction curettage), possibly reducing the rates of RPOC. RPOC. In addition, during hysteroscopy, the surgery is limited to the pregnancy implantation site, as opposed to the "global" suction curettage. This may allow for reducing the risk of postoperative intrauterine adhesions. These advantages of hysteroscopy compared to the blind suction curettage have been previously shown regarding a similar procedure, removal of RPOC by hysteroscopy compared to curettage, and nowadays it is indeed acceptable to remove RPOC primarily by hysteroscopy. Thus, it can be hypothesized that operative hysteroscopy for the management of early pregnancy loss compared with suction curettage may be associated with reduced rates of RPOC and postoperative intrauterine adhesions. On the other hand, operative hysteroscopy does have some disadvantages compared with suction curettage - it requires expensive equipment, a slightly longer operative time, and skilled surgeons. To date, few studies (mainly case series or small cohort studies) have been carried out regarding the use of hysteroscopy for surgical evacuation of early pregnancy loss. These studies found that it is an effective (feasible) and safe operation. Weinberg et al. used the hysteroscopic tissue removal device for surgical evacuation of early pregnancy loss up to 10th weeks in 10 patients. The procedure could be completed in 8 patients, and there were no significant complications. Bar-on et al. bipolar loop resectoscope in 15 women with early pregnancy loss up to 12 weeks, without short term complications. More recently, a multicenter comparative prospective study from France was published by Huchon et al. In this study, no differences were found in the rate of subsequent pregnancies. However, this study included patients who were not candidates for hysteroscopy (such as patients admitted incomplete abortion). To conclude, further comparative studies are needed to determine the benefits of operative hysteroscopy in patients with early pregnancy loss. In the present study, the investigators will perform a prospective comparison between surgical evacuation of early pregnancy loss by surgical hysteroscopy using the tissue removal device method versus the traditional suction curettage. The investigators will evaluate both the feasibility and safety (both short and long term) of the procedures, including an assessment of postoperative intrauterine adhesions.

ELIGIBILITY:
Inclusion Criteria:

1. Early pregnancy loss (miscarriage) up to 10 gestational weeks
2. Able to give informed consent, and read/write in Hebrew

Exclusion Criteria:

1. Incomplete abortion presenting as heavy vaginal bleeding and dilated cervix
2. Signs of infection and/or suspicion of septic abortion
3. Previous diagnosis of Mullerian anomalies - septate, bicornuate, unicornuate or didelphi uterus
4. Previous medical or surgical treatment in the current pregnancy
5. Previous diagnosis or past surgery for intrauterine adhesions
6. History of 2 or more prvious miscarriages
7. History of 2 or more cesarean sections
8. History of abdominal, vaginal or hysteroscopic myomectomy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Operative complications | 1 week
  Short term surgical complications including estimated blood loss > 500 ml, fluid deficit > 2500 ml, uterine perforation, re-admission, fever
Intrauterine adhesions | 6 weeks
  Assessment of intrauterine adhesions by diagnostic office hysteroscopy
Subsequent fertility | 6 months
  Rates of subsequent pregnancy

SECONDARY OUTCOMES:
Conversion from operative hysteroscopy to suction curettage | 1 day
  Inability to complete uterine evacuation by operative hysteroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Noam Smorgick, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Shamir Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Quenby S, Gallos ID, Dhillon-Smith RK, Podesek M, Stephenson MD, Fisher J, Brosens JJ, Brewin J, Ramhorst R, Lucas ES, McCoy RC, Anderson R, Daher S, Regan L, Al-Memar M, Bourne T, MacIntyre DA, Rai R, Christiansen OB, Sugiura-Ogasawara M, Odendaal J, Devall AJ, Bennett PR, Petrou S, Coomarasamy A. Miscarriage matters: the epidemiological, physical, psychological, and economic costs of early pregnancy loss. Lancet. 2021;397:1658-1667. 2. ACOG Practice Bulletin No. 200 Summary: Early Pregnancy Loss. Obstet Gynecol. 2018;132:1311-1313. 3. Shaker M, Smith A. First Trimester Miscarriage. Obstet Gynecol Clin North Am. 2022;49:623-635. 4. Upadhyay UD, Desai S, Zlidar V, Weitz TA, Grossman D, Anderson P, Taylor D. Incidence of emergency department visits and complications after abortion. Obstet Gynecol. 2015;125:175-183. 5. Paul ME, Mitchell CM, Rogers AJ, Fox MC, Lackie EG. Early surgical abortion: efficacy and safety. Am J Obstet Gynecol. 2002;187:407-11. 6. Hooker A, Fraenk D, Brölmann H, Huirne J. Prevalence of intrauterine adhesions after termination of pregnancy: a systematic review. Eur J Contracept Reprod Health Care. 2016;21:329-35. 7. Yu D, Wong YM, Cheong Y, Xia E, Li TC. Asherman syndrome--one century later. Fertil Steril. 2008;89:759-79. 8. Catena U, D'Ippolito S, Campolo F, Dinoi G, Lanzone A, Scambia G. Hysteroembryoscopy and hysteroscopic uterine evacuation of early pregnancy loss: A feasible procedure in selected cases. Facts Views Vis Obgyn. 2022;14:193-197. 9. Young S, Miller CE. Hysteroscopic resection for management of early pregnancy loss: a case report and literature review. F S Rep. 2022;3:163-167. 10. Smorgick N, Barel O, Fuchs N, Ben-Ami I, Pansky M, Vaknin Z. Hysteroscopic management of retained products of conception: meta-analysis and literature review. Eur J Obstet Gynecol Reprod Biol. 2014;173:19-22. 11. Barel O, Krakov A, Pansky M, Vaknin Z, Halperin R, Smorgick N. Intrauterine adhesions after hysteroscopic treatment for retained products of conception: what are the risk factors? Fertil Steril. 2015;103:775-9. 12. Weinberg S, Pansky M, Burshtein I, Beller U, Goldstein H, Barel O. A Pilot Study of Guided Conservative Hysteroscopic Evacuation of Early Miscarriage. J Minim Invasive Gynecol. 2021;28:1860-1867. 13. Bar-On S, Berkovitz Shperling R, Cohen A, Akdam A, Michaan N, Levin I, Rattan G, Tzur Y. Primary Resectoscopic Treatment of First-Trimester Miscarriage. J Obstet Gynaecol Can. 2023:102327. 14. Huchon C, Drioueche H, Koskas M, Agostini A, Bauville E, Bourdel N, Fernandez H, Fritel X, Graesslin O, Legendre G, Lucot JP, Panel P, Raiffort C, Giraudet G, Bussières L, Fauconnier A. Operative Hysteroscopy vs Vacuum Aspiration for Incomplete Spontaneous Abortion: A Randomized Clinical Trial. JAMA. 2023;329:1197-1205.